CLINICAL TRIAL: NCT07130565
Title: Pan-Amyloid PET/CT in Various Amyloid-Related Disease
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Prof., Tianjin Medical University
Other Study IDs: TJMUGH-11
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Amyloid; Cardiac Amyloidosis; Amyloidosis
Keywords: PET/CT; MRI; Pan-Amyloid
MeSH Terms: conditions — Alzheimer Disease; Amyloid Neuropathies, Familial; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: Each subject receive a single intravenous injection of 18F-92/AV45/TPZA/FT8, 11CPIB and undergo PET/CT or MRI imaging within the specificed time.
  Interventions: Diagnostic Test: 18F-92/AV45/TPZA/FT8, 11CPIB

INTERVENTIONS:
Diagnostic Test: 18F-92/AV45/TPZA/FT8, 11CPIB — Each subject receive a single intravenous injection of 18F-92/AV45/TPZA/FT8, 11C-PIB and undergo PET/CT or MRI imaging within the specificed time.

SUMMARY:
To evaluate the potential usefulness of 18F-92/AV45/TPZA/FT8, 11C-PIB positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various Pan-Amyloid-related disease patients.

DETAILED DESCRIPTION:
Subjects with various Pan-Amyloid-related disease patients underwent 18F-92/AV45TPZA/FT8, 11C-PIB PET/CT either for an initial assessment or for recurrence detection. Lesions uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-92/AV45TPZA/FT8, 11C-PIB PET/CT were calculated.

ELIGIBILITY:
Inclusion Criteria:

- (i) adult patients (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated cardiac amyloidosis (supporting evidence may include MRI, CT, serum markers and pathology report); (iii) patients who had scheduled Pan-Amyloid PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

- (i) patients with non-CA lesions; (ii) patients with pregnancy; (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (i) adult patients (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated CA (supporting evidence may include MRI, CT, tumor markers and pathology report); (iii) patients who had scheduled amyloid PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of 18F-92/AV45/TPZA/FT8, 11C-PIB for each target lesion of subject or suspected Pan-Amyloid related diseases.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of Pan-Amyloid PET/CT were calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No